CLINICAL TRIAL: NCT05948592
Title: A Phase 2 CT to Evaluate the Safety and Efficacy of Topical Administration of Bacteriophage Therapy TP-102 in Patients With DFI
Brief Title: Bacteriophage Therapy TP-102 in Patients With Diabetic Foot Infection
Acronym: REVERSE2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technophage, SA (Industry)
Collaborators: VectorB2B (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TP-102_102
Record Dates: First submitted 2023-06-15; First posted 2023-07-17 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Foot Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TP-102 (Experimental): Patients will be randomly assigned in a 1:1 ratio to one of two treatment arms at Day 1. The wound standard of care (SoC) procedures shall be in accordance to each sites normal DFI routine.
  Interventions: Biological: TP-102
- Placebo (Placebo Comparator): Patients will be randomly assigned in a 1:1 ratio to one of two treatment arms at Day 1. The wound standard of care (SoC) procedures shall be in accordance to each sites normal DFI routine.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: TP-102 — Patients randomised to TP-102 will receive 1 (one) mL of IP solution, applied topically per cm3 of target ulcer. The titre of each bacteriophage in TP-102 is 1x109 PFU/mL (>1x108 PFU/mL and <1x1010 PFU/mL). All patients randomised to TP-102 will receive the same concentration per mL. TP-102 will be applied to the target ulcer using a syringe without a needle. The volume of TP-102 to be administered will be determined from the wound volume assessment at the previous visit through an automated wound measurement system (Silhouette), except on the first day of treatment where the amount applied will be determined based on the wound volume determined at that time using the automated wound measurement system (Silhouette).
  Arms: TP-102
Other: Placebo — Patients randomised to placebo, the volume calculated to be administered will be determined from the wound volume assessment at the previous visit through an automated wound measurement system (Silhouette), except on the first day of treatment where the amount applied will be determined based on the wound volume determined at that time using the automated wound measurement system (Silhouette).
  Arms: Placebo

SUMMARY:
TP-102 is a novel bacteriophage cocktail comprised of 5 (five) lytic bacteriophages against Staphylococcus aureus, Pseudomonas aeruginosa, and Acinetobacter baumannii. TP-102 is being developed for topical treatment of patients with wound infections including chronic ulcers; applied every other day (three times weekly (TIW)).

DETAILED DESCRIPTION:
This is a Phase 2b, double-blinded, randomised, placebo-controlled multicenter study to determine the safety and efficacy of TP-102, in patients with diabetic foot infection.

Eighty (80) patients with an infected diabetic foot ulcer and with at least one target bacterial strain (Pseudomonas aeruginosa, Staphylococcus aureus or Acinetobacter baumannii) susceptible to TP-102.

Patients will be randomised to receive TP-102 or placebo, in a 1:1 ratio. Patients will be treated with 1 (one) mL of IP/ Placebo solution applied topically per cm3 of target ulcer. Patients will be treated with a total of 12 treatments in 28 days (+3 days) with at least one day of interval in between the days of treatment (no consecutive days of treatment are allowed) and a maximum of 3 (three) days without treatment.

The titre of each bacteriophage in TP-102 is 1x109 (>1x108 and < 1x1010) plaque forming units per milliliter (PFU/mL).

Assessments for efficacy and safety will include concomitant medications and AEs, local tolerability, clinical laboratory tests, vital signs, physical examination, wound biopsy/swab to determine the presence, speciation and TP-102 sensitivity of bacteria and target ulcer assessment.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years old;
* Established diagnosis of Diabetes Mellitus (type I or II);
* Glycosylated hemoglobin (HbA1c) value < 12.0%;
* Designated foot infection meets the following criteria:
* Present for at least 3 weeks;
* Below-ankle, full-thickness, cutaneous ulcer;
* Wound area (after debridement, if applicable) 1 to 20.0 cm2;
* PEDIS infection grade 2 or 3;
* PEDIS perfusion grade 1 or 2;
* PEDIS depth grade 1 or 2 (grade 3 at the discretion of the investigator e.g. if they have received appropriate surgical treatment to remove infected bones).
* Diabetic foot infection with at least one target bacterial strain (Pseudomonas aeruginosa, Staphylococcus aureus or Acinetobacter baumannii), susceptible to the TP-102 bacteriophage cocktail, as assessed from wound cultures;
* Patients of suitable physical and mental health as determined by the Investigator on the basis of medical history and general physical examination;
* Patients of childbearing potential must have a negative serum pregnancy test at screening;
* ICF signed voluntarily before any study-related procedure is performed, indicating that the patient understands the purpose of, and procedures required in the study and is willing to participate in the study.

Exclusion Criteria:

* Infected study ulcer less than 2 cm away from other ulcers, in the case of multiple ulcers;
* Patient receiving hyperbaric oxygen therapy (HBOT), negative pressure wound therapy (NPWT), bioengineering skin (BES) substitutes and/or growth factors;
* Patient which, in the opinion of the investigator, may not comply with study related procedures;
* Presence of active malignant or benign tumors of any kind, (with exception to nonmelanoma skin cancer as per investigator's discretion);
* Being pregnant or breastfeeding;
* Currently participating in another clinical trial or having participated in a previous clinical trial with receipt of an investigational product within 30 days of the first administration of IP;
* A condition that, in the opinion of the Investigator, could compromise the well-being of the patient or course of the study, or prevent the patient from meeting or performing any study requirements;
* Participants with hypersensitivity to any component of investigational products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
1. Number and percentage of treatment emergent adverse events (TEAEs) | From baseline to EOT, aproximately 12 weeks
  See above
2. Mean DFUWI score (total AUC) for TP-102 versus Placebo | From baseline to EOT, , aproximately 12 weeks
  See above
3. Percentage of patients that achieve a 50% reduction in wound surface area by week 4 | Week 4

SECONDARY OUTCOMES:
1. Change in mean CRP/ESR/PCT/WCC value for TP-102 versus Placebo | From baseline to EOT, , aproximately 12 weeks
2. Percentage of patients with a value over clinical diagnostic cut-off for DFI for CRP/ESR/PCT/WCC | Baseline to EOT, , aproximately 12 weeks
3. Percentage eradication of TP-102 susceptible strains for TP-102 versus Placebo at EOT; | EOT, , aproximately 12 weeks
4. Percentage of patients with target strain not-susceptible to TP-102 for TP-102 versus Placebo at EOT; | EOT, , aproximately 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Arsule, Principal Investigator — Shree Siddhi Vinayal Hospital; Yalamanchi Rao, Principal Investigator — Yalamanchi Hospitals & Research Centers Pvt. Ltd; Senthil Kumar, Principal Investigator — MV Hospital for Diabetes Pvt. Ltd; Aman Khanna, Principal Investigator — Aman Hospital & Research Centre; Mohammad Qureshi, Principal Investigator — Crescent Hospital & Heart Centre; Parikh Niranjan, Principal Investigator — Parikh Multispeciality Healthcare Pvt. Ltd; Sanjay Kala, Principal Investigator — GSVM Medical College; Vikas Matai, Principal Investigator — Jupiter Hospital & Research Centre; Stan Mathis, PI, Principal Investigator — Clemente Clinical Research; Abdul Moosa, PI, Principal Investigator — Tranquil Clinical Research
Locations (10):
- United States (2):
  - Clemente Clinical Research, Los Angeles, California
  - Tranquil Clinical Research, Webster, Texas
- India (8):
  - MV Hospital for Diabetes Pvt. Ltd, Chennai
  - GSVM Medical College, Kanpur
  - Crescent Hospital & Heart Centre, Nagpur
  - Shree Siddhi Vinayak Hospital, Nashik
  - Jupiter Hospital & Research Center, Vadodara
  - Parikh Multispeciality Healthcare Pvt. Ltd, Vadodara
  - Aman Hospital & Research Centre, Vadodara
  - Yalamanchi Hospitals & Research Centers Pvt. Ltd, Vijayawada

IPD SHARING:
Plan to Share IPD: No